CLINICAL TRIAL: NCT02418637
Title: Worksite Screening for Cardiovascular Risk Factors Among Migrant Agricultural Workers
Brief Title: Pilot Study Testing Feasibility of Health Screening at Farm Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, M. Hassan Murad, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-000647
Record Dates: First submitted 2015-04-06; First posted 2015-04-16 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Screening; Hyperlipidemia Screening; Hypertension Screening
Keywords: worksite; screen; migrant; agricultural; worker; hypertension; Hyperlipidemia; diabetes; feasibility
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Farm workers (Experimental): This is a one arm intervention including farm workers and owners
  Interventions: Other: Worksite screening for DM, HTN and hyperlipidemia

INTERVENTIONS:
Other: Worksite screening for DM, HTN and hyperlipidemia — Six monthly visits to worksite to perform screenings

SUMMARY:
Test the feasibility of performing worksite screening of Hypertension, Diabetes and Hyperlipidemia for six months

DETAILED DESCRIPTION:
The investigators will be visiting farmers at the worksite monthly for six month and perform cardiovascular risk factors screening: blood pressure, blood glucose, glycosylated hemoglobin and cholesterol.

At the end of this intervention, the investigators will test the feasibility of this approach among this specific population through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* agricultural workers and farm owners

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility (Likert scale) | After six months of the intervention, the outcome will be assessed on the last site visit via questionnaire
  On a likert scale, the investigators will test the applicability, acceptance and convenience of this screening approach among this agricultural workers population

CONTACTS AND LOCATIONS:
Overall Officials: M Murad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Rajjo T, Mohammed K, Rho J, Murad MH. On-the-farm cardiovascular risk screening among migrant agricultural workers in Southeast Minnesota: a pilot prospective study. BMJ Open. 2018 Jul 30;8(7):e019547. doi: 10.1136/bmjopen-2017-019547. PMID 30061429